CLINICAL TRIAL: NCT01220401
Title: Efficacy of a Brief Nightmare Treatment for Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tulsa (Other)
Responsible Party: Principal Investigator, Joanne Davis, PI, University of Tulsa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TU1107
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Sleep Disorders; PTSD; Suicide
Keywords: Nightmare; PTSD; Posttraumatic stress disorder; Suicide; Exposure Relaxation Rescription Therapy; Sleep
MeSH Terms: conditions — Sleep Wake Disorders; Stress Disorders, Post-Traumatic; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ERRT-M (Experimental): Exposure, Relaxation, and Rescripting Therapy for military populations. 4 sessions.
  Interventions: Behavioral: exposure, relaxation, and rescription therapy

INTERVENTIONS:
Behavioral: exposure, relaxation, and rescription therapy — veterans reporting chronic nightmares at least once per week for the past month who consent to participate will attend four consecutive weekly sessions lasting approximately two hours each. Participants will log their sleep events and associated symptoms (i.e. PTSD, depression, etc.)

SUMMARY:
The purpose of this study is to find out what effects Exposure, Rescripting, and Relaxation Therapy (ERRT) has on nightmares and associated problems in veterans.

DETAILED DESCRIPTION:
The purpose of the proposed pilot study is to extend previous findings regarding the impact of a brief cognitive behavioral treatment for chronic nightmares by examining the emotional, cognitive, behavioral, and health-related changes following treatment. Experiencing a traumatic event may initiate or exacerbate the occurrence of nightmares. Indeed, sleep disturbance, including nightmares, is considered a hallmark of posttraumatic stress disorder (PTSD). Nightmares have been related to a variety of factors including stress, medications, trauma, and substance use. Among veterans, especially combat veterans or those reporting sexual assaults, symptoms of traumatic stress and nightmares are extremely common. Few studies have investigated the efficacy of nightmare treatment in a veteran population, and the impact of nightmare treatment on suicidal ideation has never been assessed.

Imagery Rehearsal Treatment (IRT) has received increased attention in the past decade for use with chronic nightmares. Studies suggest that the treatment is promising for the reduction of frequency and intensity of chronic nightmares in trauma exposed persons and may have a generalized impact on symptoms of posttraumatic stress disorder and depression and quality/quantity of sleep, although there is mixed evidence for sleep improvement among veterans. The principal investigator has completed two randomized controlled trials of a modified version of IRT, Exposure, Rescripting, and Relaxation Treatment (ERRT) and is currently conducting a third randomized controlled trial (Davis, 2008; Davis & Wright, 2007). The current randomized controlled trial is comparing ERRT to an active treatment (relaxation). Results demonstrated positive treatment response. Although these trials have included some veteran participants, veterans have not been studied as a group using this protocol. The purpose of this prospective study is to conduct a pre- and post-treatment comparison of suicidal ideation and posttraumatic, depressive, and health symptoms in a single group of veterans.

ELIGIBILITY:
Inclusion Criteria: veteran/military, 18+ years old, english proficiency, nightmares once per week, exposure to a criterion A traumatic event -

Exclusion Criteria: under 18, psychotic illness, mental retardation, imminent suicidal intent

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noelle Balliett, MA, Principal Investigator — The University of Tulsa
Locations (1):
- The University of Tulsa, Tulsa, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ERRT-M
Started | 21
Completed | 18
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | ERRT-M
Number analyzed (Participants) | 21
Age, Customized [Mean (Standard Deviation); unit: years] | 56.6 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 6
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Nights With Nightmares
Description: This fill-in-the-blank variable assesses the number of nights the individual experienced nightmares in the past week (range = 0 - 7 nights). Higher values indicate more nights with nightmares (worse outcome).
Time Frame: pre, one week, two months
Measure: Mean (Standard Deviation); unit: nights/week
Groups:
- ERRT-M: Exposure, Relaxation, and Rescripting Therapy for military populations. 4 sessions.
  exposure, relaxation, and rescription therapy: veterans reporting chronic nightmares at least once per week for the past month who consent to participate will attend four consecutive weekly sessions lasting approximately two hours each. Treatment consists of psychoeducation, relaxation techniques, mindfulness, exposure to nightmare content, and rescription of nightmare to make it less distressing.
  Participants will log their sleep events and associated symptoms (i.e. PTSD, depression, etc.)
Arm/Group | ERRT-M
Number analyzed (Participants) | 18
nights/week
  Baseline Nights with Nightmares | 2.61 (1.79)
  1-week Nights with Nightmare | .83 (1.20)
  2-month Nights with Nightmare | 0.97 (1.23)

2. Primary Outcome: Clinician Administered PTSD Scale
Description: This semi-structured clinical interview assesses each of 17 DSM-IV-TR criteria for PTSD utilizing separate queries for frequency and severity on a 5-point scale (0 - 4). This study utilized the "FI/I2" rule, where frequency ratings of one or more and intensity ratings of two or more must be present in order for a symptom to count towards diagnosis.
  Total scores are comprised of the three factors (reexperiencing, avoidance, and hyperarousal), with 136 being the maximum. 0-19 = asymptomatic or few symptoms. 20-39 = mild PTSD, subthreshold. 40-59 = moderate PTSD at threshold. 60-79 = severe PTSD. 80+ = extreme PTSD.
Time Frame: pre, one week, two months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ERRT-M
Number analyzed (Participants) | 18
units on a scale
  Baseline TOTAL PTSD | 50.72 (24.60)
  1-week TOTAL PTSD | 46.44 (27.62)
  2-month TOTAL PTSD | 43.00 (23.10)

3. Secondary Outcome: Beck Depression Inventory
Description: This 21-item, self-report measure was designed to assess the severity of depression among adults. Responses on a Likert-type scale range from 0 - 3, and scores may be summed to derive a total score (0-63), with higher scores indicating more depressive symptoms. Scores of 18 and above have been suggested to reliably identify depressed patients.
Time Frame: Baseline, 1 week, 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ERRT-M
Number analyzed (Participants) | 18
units on a scale
  Baseline Depression | 27.61 (11.72)
  1-week Depression | 18.94 (8.90)
  2-month Depression | 22.11 (11.11)

4. Primary Outcome: Past Week Nightmare Frequency
Description: This fill-in-the-blank variable assesses the number of nightmares experienced in the past week (range = 0 - X nightmares). Higher values indicate more nightmares (worse outcome).
Time Frame: pre, one week, two months
Measure: Mean (Standard Deviation); unit: nightmares/week
Arm/Group | ERRT-M
Number analyzed (Participants) | 18
nightmares/week
  Baseline Nightmare Frequency (# in past week) | 2.97 (1.78)
  1 Week Nightmare Frequency (# in past week) | 1.17 (1.48)
  2 Month Nightmare Frequency (# in past week) | 1.03 (1.30)

ADVERSE EVENTS:
Arm/Group | ERRT-M
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No